CLINICAL TRIAL: NCT05762926
Title: Non-invasive Brain Stimulation by Transcranial Pulse Stimulation as a Coadjunctive Treatment in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 54939622.1.0000.0068
Record Dates: First submitted 2022-07-20; First posted 2023-03-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Transcranial Magnetic Stimulation; Extracorporeal Shockwave Therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double (Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental: Neuronavigation system guided halocranial application of focused sound wave pulses, using the Storz Neurolith™ equipment.
  Interventions: Other: Transcranial pulse stimulation (TPS)
- Active Comparator (Active Comparator): Neuronavigation system guided halocranial application without sound waves pulses, using the Storz Neurolith™ sham equipment, prepared to block the sound waves.
  Interventions: Other: Transcranial pulse stimulation (TPS)

INTERVENTIONS:
Other: Transcranial pulse stimulation (TPS) — Clinical treatment consists in ten sessions of neuronavigation system guided halocranial application of 6000 focused sound wave pulses, with energy flux density of 0.25 mJ/mm2, depth of focus of 5 cm and useful energy between 4 to 6 cm, frequency of 4 Hz, total energy applied will be 50 Joules, for it will be used the Storz Neurolith™ equipment.

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial; that will evaluate the effectiveness of the use of transcranial pulse stimulation in people living with Alzheimer's disease, coming from the Institute of Psychiatry (IPQ) of the Hospital das Clinicas, Faculty of Medicine, University of São Paulo, and the Institute of Physical Medicine and Rehabilitation (IMREA) at the Hospital das Clínicas, Faculty of Medicine, University of São Paulo.

Participants will be classified according to the stage of Alzheimer's disease, determined by a psychiatrist and neuropsychologists. A total of 50 volunteers will be randomized blindly. In addition to evaluating the clinical course and imaging examination, the use of scales that assess functional and cognitive disability will be used for the recruitment of volunteers. Volunteers will be randomized into two study groups, and will receive the intervention that will consist of ten sessions, held twice a week. The Storz Neurolith™ equipment (Storz Medical, Tagerwillen, Switzerland) will be used to administer transcranial pulse stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have Alzheimer's disease will be selected;
* Are aged ≥50 years;
* Medical assistance provided by the psychiatry service at IPQ;
* Who agree to participate after consent via the Informed Consent Term .

Exclusion Criteria:

* Make regular use of anticoagulants;
* Has skullcap failure, craniectomy without cranioplasty;
* Have a diagnosis of brain neoplasms or any type of nodule in the brain region;
* Have recent brain bleeds or a diagnosis of cerebral arteriovenous malformation;
* Be diagnosed with a type of dementia other than Alzheimer's;
* Have Mild Cognitive Impairment of the Elderly (MCI);
* Have clinical changes that put the test at risk, such as severe cardiorespiratory disorders;
* Has a severe cognitive disorder that makes it impossible to apply therapy or questionnaires;
* It is clinically or socially impossible for the patient to attend IMREA for applications twice a week during the study period;
* Those who disagree to participate after consent via the Informed Consent Term .

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 50 Years and older (Adult, Older Adult)
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Cognitive Functions | Baseline and up to one, three, six and twelve months from intervention
  Cognitive functions, using Alzheimer's Disease Assessment Scale (ADAS-Cog)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Medicina Física e Reabilitação, Hospital das Clínicas, Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) may be shared in the future under suitable request and justification to principal investigator.